CLINICAL TRIAL: NCT01463904
Title: Single-Anastomosis Duodeno-Ileal Bypass With Sleeve Gastrectomy (SADI-S) for the Treatment of Morbid Obesity and Its Metabolic Complications
Acronym: SADI-S 250
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Andres Sanchez-Pernaute, MD, PhD, Hospital San Carlos, Madrid
Other Study IDs: FMMA-08 Sánchez-Pernaute
Record Dates: First submitted 2011-10-31; First posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Morbid Obesity; Diabetes
Keywords: Morbid obesity; duodenal switch; diabetes; decrease in cardiac risk; remission of T2DM
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of subcutaneous and visceral fat, and samples of liver tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Morbid obese, diabetics: Patients with morbid obesity or severe metabolic disease
  Interventions: Procedure: SADI-S 250

INTERVENTIONS:
Procedure: SADI-S 250 — Single-Anastomosis Duodeno-Ileal bypass with Sleeve gastrectomy

SUMMARY:
Single-Anastomosis Duodeno-Ileal Bypass with Sleeve Gastrectomy is a modified and simplified duodenal switch. It is performed on morbid obese patients and severe T2DM patients with obesity, and a proper weight loss is expected as well as a decrease in the cardiac risk and a remission of T2DM. A lower complication rate than for duodenal switch is expected.

DETAILED DESCRIPTION:
A sleeve gastrectomy over a wide bougie is performed. Then the proximal duodenum is divided and anastomosed to the ileum 250 cm from the cecum.

The preoperative studies and postoperative follow up is similar to those performed before and after other bariatric procedures.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 with T2DM or BMI > 40

Exclusion Criteria:

* Oncologic patients, alcoholic patients, mentally retarded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Morbid obesity patients and patients with obesity and T2DM
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-07 (Actual); Study Completion 2015-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain